CLINICAL TRIAL: NCT06041555
Title: MRI Guided Radiotherapy and Radiobiological Data: the ISRAR Database (Irm Sequences for Radiobiological Adaptative Radiotherapy)
Acronym: ISRAR
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0298; 2023-A01124-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Glioblastoma; Head and Neck Cancer; Kidney Cancer; Cervix Cancer
Keywords: LINAC; MRI; Radiotherapy; Mapping; Hypoxia; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Glioblastoma; Head and Neck Neoplasms; Kidney Neoplasms; Uterine Cervical Neoplasms; Hypoxia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ISRAR Cohort: All patient treated with the LINAC UNITY MRI radioguided radiotherapy for a prostate, kidney cancer, cervix, head and neck cancer or glioblastoma.
  Interventions: Other: 3 MRI sequences (T2*, IVIM and Multi Echo-Gradient), without injection, are performed

INTERVENTIONS:
Other: 3 MRI sequences (T2*, IVIM and Multi Echo-Gradient), without injection, are performed — Generate 3D maps of intra-tumoral hypoxia and characterize their evolution during treatment thanks to the establishment of a prospective database of MRI sequences

SUMMARY:
The MRI linac Unity is a major technological evolution in radiotherapy combining a linear accelerator with a 1.5T MRI (radiological quality). It allows to target the target volume more precisely and to adapt the daily dose distribution according to variations in the position and volume of the tumor, critical organs and the tumor response. In many studies conducted in radiology, the analysis of specific MRI sequences, particularly in radiomics, aims to characterize tumors and their sensitivity to treatment. Initial data show that in radiotherapy, it would eventually be possible to characterize the radiosensitivity of healthy and tumorous tissues. With linac 1.5T MRI, the performance of selected MRI sequences, at each session, could make it possible to identify different levels of radiosensitivity within the tumour. The reproduction of these sequences on a daily basis could make it possible to follow the variations in radiosensitivity during the treatment. The final objectives would be: 1- to adapt the doses of radiotherapy to each session with a modulation of the dose according to the daily level of intra-tumor radiosensitivity, 2- to develop Artificial Intelligence (AI) tools allowing an analysis sequences and the generation of 3D maps of intra-tumor radiosensitivity, fast and suitable for carrying out a radiotherapy session.

A first work carried out in collaboration with the CREATIS lab of the University Claude Bernard Lyon 1 (UCBL1) made it possible to generate maps of tissue oxygenation from sequences produced on the MRI linac Unity of the Hospices Civils de Lyon (T2* , IVIM, Carto T2 Multi Echo-Gradient). Hypoxia is known to be the first factor of tumor resistance to irradiation. A research program is structured in collaboration with UCBL1 in order to develop radiobiological adaptive radiotherapy approaches, based on 3D maps of intra-tumoral hypoxia and their variation during treatment. Several tumor locations were selected because of the preponderant place of MRI in tumor characterization: prostate, cervix, kidney, ENT and glioblastoma. Hypoxia is not the only factor of radioresistance. Changes in the microenvironment could also impact the sensitivity of tumor cells. The program will therefore also aim to optimize the maps initially based on hypoxia, by identifying other relevant factors to be taken into account to define intra-tumor sensitivity.

DETAILED DESCRIPTION:
The MRI linac Unity is a major technological evolution in radiotherapy combining a linear accelerator with a 1.5T MRI (radiological quality). It allows to target the target volume more precisely and to adapt the daily dose distribution according to variations in the position and volume of the tumor, critical organs and the tumor response. In many studies conducted in radiology, the analysis of specific MRI sequences, particularly in radiomics, aims to characterize tumors and their sensitivity to treatment. Initial data show that in radiotherapy, it would eventually be possible to characterize the radiosensitivity of healthy and tumorous tissues. With linac 1.5T MRI, the performance of selected MRI sequences, at each session, could make it possible to identify different levels of radiosensitivity within the tumour. The reproduction of these sequences on a daily basis could make it possible to follow the variations in radiosensitivity during the treatment. The final objectives would be: 1- to adapt the doses of radiotherapy to each session with a modulation of the dose according to the daily level of intra-tumor radiosensitivity, 2- to develop Artificial Intelligence (AI) tools allowing an analysis sequences and the generation of 3D maps of intra-tumor radiosensitivity, fast and suitable for carrying out a radiotherapy session.

A first work carried out in collaboration with the CREATIS lab of the University Claude Bernard Lyon 1 (UCBL1) made it possible to generate maps of tissue oxygenation from sequences produced on the MRI linac Unity of the Hospices Civils de Lyon (T2* , IVIM, Carto T2 Multi Echo-Gradient). Hypoxia is known to be the first factor of tumor resistance to irradiation. A research program is structured in collaboration with UCBL1 in order to develop radiobiological adaptive radiotherapy approaches, based on 3D maps of intra-tumoral hypoxia and their variation during treatment. Several tumor locations were selected because of the preponderant place of MRI in tumor characterization: prostate, cervix, kidney, ENT and glioblastoma. Hypoxia is not the only factor of radioresistance. Changes in the microenvironment could also impact the sensitivity of tumor cells. The program will therefore also aim to optimize the maps initially based on hypoxia, by identifying other relevant factors to be taken into account to define intra-tumor sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 18years old or older
* diagnosed with prostate, kidney, cervix, head and neck cancer or glioblastoma
* indication of external radiotherapy
* treated with the Linac UNITY MRI guided radiotherapy at the centre hospitalier Lyon Sud des Hospices Civils de Lyon
* agreement of the patient to participate
* affiliated to a social security system

Exclusion Criteria:

patient unable to keep a lying position during all the procedure

* patient under law restriction
* pregnant women or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient treated with the LINAC UNITY MRI radioguided radiotherapy for a prostate, kidney cancer, cervix, head and neck cancer or glioblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Hypoxia mapping | At the end of the sequence of treatment of each patient, that is 13 weeks after the beginning of the treatment
  Generate 3D maps of intra-tumoral hypoxia and characterize their evolution during treatment thanks to the establishment of a prospective database of MRI sequences

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud/ service de Radiothérapie Oncologie, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided